CLINICAL TRIAL: NCT07380971
Title: From Scientific Evidence to Practice: Developing a Comprehensive Exercise Service for Breast Cancer Process
Brief Title: Developing a Comprehensive Exercise Service for Breast Cancer Process
Status: Recruiting | Type: Observational
Sponsor: GO fit Lab- Ingesport (Network)
Responsible Party: Sponsor
Other Study IDs: Moving Together
Record Dates: First submitted 2025-11-17; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Exercise; Physical activity; Complementary Therapy; Personalized Exercise Program; Implementation Science; Hospital-based Exercise; Cancer Rehabilitation
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Supervised In-Person Exercise Group: Participants in this group engage in supervised, in-person exercise sessions at the GO fit Vallehermoso center.
  Interventions: Other: Supervised in-person exercise training
- Supervised Online Exercise Group: Participants in this group follow the same structured exercise program as the in-person group but attend sessions via live video conferencing.
  Interventions: Other: Supervised Online Exercise Training
- Autonomous Home-Based Exercise Group: Participants receive structured exercise guidelines to follow independently at home.
  Interventions: Other: Home-Based Autonomous Exercise Program
- Autonomous Gym-Based Exercise Group: Participants follow individualized exercise guidelines at gym, using gym equipment for strength and aerobic training.
  Interventions: Other: Gym-Based Autonomous Exercise Program
- Control Group (Usual Care): Participants in this group do not engage in any of the structured exercise programs but continue with their standard medical care and follow-up.
  Interventions: Other: Usual Care Without Structured Exercise

INTERVENTIONS:
Other: Supervised in-person exercise training — Participants attend 60-minute, twice-weekly exercise sessions at GO fit Vallehermoso. Sessions include warm-up, aerobic and resistance training, and cool-down. Exercises are tailored to the patient's treatment phase (pre-surgery, during chemotherapy/radiotherapy, or survivorship) and adjusted based on symptoms like fatigue or pain. Heart rate is monitored in real time. Groups are formed by treatment phase and physical capacity to ensure safety and personalization.
  Groups: Supervised In-Person Exercise Group
Other: Supervised Online Exercise Training — Participants follow the same structure as the in-person group but attend sessions via live video conferencing. They receive equipment and training on using the MYZONE app for heart rate monitoring. Sessions are interactive, allowing real-time feedback and social support. This option is designed for patients with mobility, time, or travel limitations.
  Groups: Supervised Online Exercise Group
Other: Home-Based Autonomous Exercise Program — Participants receive structured exercise guidelines to follow independently at home. Programs include aerobic and strength exercises using bodyweight or household items, with three levels of progression. Training is recommended 1-3 times per week. Participants track activity using a diary and smartphone accelerometer. Programs are adapted to treatment phase and personal capacity.
  Groups: Autonomous Home-Based Exercise Group
Other: Gym-Based Autonomous Exercise Program — Participants follow individualized exercise guidelines at the gym, using gym equipment for strength and aerobic training. The program is self-directed but based on the same structure and progression as supervised programs. Activity is tracked via accelerometers and exercise logs. Participants choose this option based on preference and access to gym facilities.
  Groups: Autonomous Gym-Based Exercise Group
Other: Usual Care Without Structured Exercise — Participants in this group do not receive any structured exercise intervention. They continue with standard medical care and follow-up as prescribed by their oncology team. They undergo the same clinical, physical, and psychological assessments as the intervention groups to allow for comparison of outcomes.
  Groups: Control Group (Usual Care)

SUMMARY:
"Moving Together" (Juntas en Movimiento) is a hospital-based, comprehensive, and personalized exercise service designed for women diagnosed with breast cancer. This implementation study aims to evaluate the feasibility, safety, and impact of integrating a free, tailored exercise program into routine clinical care at Hospital Clínico San Carlos in Madrid, Spain.

The program offers multiple participation options-supervised in-person, supervised online, autonomous at home, or autonomous at a fitness center-allowing patients to choose based on their preferences, limitations, and treatment phase (pre-surgery, during chemotherapy/radiotherapy, or survivorship). All exercise options are adapted to individual needs and include aerobic and resistance training components.

The study uses a real-world implementation science approach, guided by the Consolidated Framework for Implementation Research (CFIR), to assess clinical, physical, and psychological outcomes such as quality of life, cardiorespiratory fitness, muscle strength, body composition, and adherence to physical activity. Data are collected through clinical records, physical assessments, validated questionnaires, and wearable technology.

This pioneering initiative in Spain seeks to establish exercise as a standard complementary therapy in oncology care, bridging the gap between scientific evidence and clinical practice, and promoting long-term health and well-being in breast cancer patients.

DETAILED DESCRIPTION:
"Moving Together" (Juntas en Movimiento) is an implementation research project that evaluates the integration of a comprehensive, free, and personalized exercise service into the clinical care of women with breast cancer. The service is embedded within the Breast Unit of Hospital Clínico San Carlos (Madrid, Spain) and is developed in collaboration with King Juan Carlos University and GO fit Vallehermoso.

The program is designed to be inclusive and adaptable, offering four participation modalities:

* Supervised in-person sessions at a fitness center.
* Supervised online sessions via video conferencing.
* Autonomous home-based training with structured guidelines.
* Autonomous training at a gym with tailored routines.

Patients can join the program at any stage of their cancer journey-before surgery, during chemotherapy or radiotherapy, or in the survivorship phase. The exercise protocols are adapted to each phase and personalized based on clinical status, physical capacity, preferences, and daily symptoms. Supervised sessions include real-time heart rate monitoring and are delivered in small groups to foster social support.

The implementation follows the CFIR model, analyzing internal and external factors that influence adoption, sustainability, and scalability. The program is supported by interdisciplinary collaboration among oncologists, gynecologists, exercise scientists, and clinical staff. Healthcare professionals receive specific training to promote exercise as part of cancer care.

Assessments include:

* Clinical data (tumor type/stage, treatments, biomarkers).
* Physical evaluations (body composition, strength, flexibility, balance, cardiorespiratory fitness).
* Psychological and behavioral measures (quality of life, physical activity levels, perceived barriers/benefits, adherence).

Data are collected using REDCap and wearable devices (e.g., accelerometers, heart rate monitors). Behavioral change strategies, including the COM-B model and the PADEX checklist, are applied to enhance motivation, self-efficacy, and long-term adherence.

The program also fosters a supportive community through workshops, group sessions, and family-inclusive events. It aims to humanize care, empower patients, and create a sustainable model for integrating exercise into oncology services.

This initiative not only improves patient outcomes but also creates a real-world research platform to explore the effects of exercise across different cancer stages and patient profiles. Future randomized controlled trials will be embedded within the service to refine exercise prescriptions and optimize clinical impact.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older.
* Diagnosed with any type and stage of breast cancer.
* Receiving care at Hospital Clínico San Carlos (Madrid, Spain).
* Willing and able to provide informed consent.
* Eligible to participate in physical activity based on clinical evaluation.

Exclusion Criteria:

* Medical contraindications to physical exercise.
* Severe uncontrolled conditions (whether related to cancer treatment or not).
* Diagnosis of recurrent breast cancer.
* Refusal or inability to sign the informed consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years or older diagnosed with any type and stage of breast cancer, receiving care at Hospital Clínico San Carlos (Madrid, Spain). Participants may be at any phase of treatment (pre-surgery, during chemotherapy or radiotherapy, or in the survivorship phase). The study includes a diverse population with varying clinical profiles, physical capacities, and personal circumstances. The exercise program is inclusive and personalized, allowing participation regardless of treatment type or modality, as long as there are no medical contraindications to physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life (HRQoL) measured by the EORTC QLQ-C30 | Baseline, 4 months, 8 months, and 12 months after enrollment
  Health-related quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). This instrument includes functional scales, symptom scales, and a global health status scale, all scored from 0 to 100. Higher scores on functional and global health scales indicate better quality of life, whereas higher scores on symptom scales indicate greater symptom burden. The outcome is the change in QLQ-C30 scores from baseline to 4, 8, and 12 months.
Change in Health-Related Quality of Life (HRQoL) measured by the EORTC QLQ-BR42 | Baseline, 4 months, 8 months, and 12 months after enrollment
  HRQoL specific to breast cancer will be assessed using the EORTC Breast Cancer-Specific Module (QLQ-BR42). This questionnaire produces scores ranging from 0 to 100. Higher symptom scores indicate worse symptom burden.

SECONDARY OUTCOMES:
Change in VO2 peak during the cardiorespiratory fitness test | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Measured using a submaximal test to estimate VO₂peak before and after the exercise program.
Change in heart rate response during the cardiorrespiaroty test | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Measured using a submaximal test to record heart rate response before and after te exercise program.
Change in blood lactate concentration during the cardiorespiratory fitness test | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Measured using a submaximal test to measure blood lactate concentration before and after the exercise program.
Change in physical activity levels | Continuous monitoring; summarized at baseline, 6 and 12 months
  Measured using the IPAQ-SF questionnaire and daily step counts via smartphone apps or accelerometers.
Change in Weight | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Body weight measured using a calibrated digital scale before and after the intervention.
Change in Musculoskeletal Mass | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Musculoskeletal mass assessed using bioelectrical impedance analysis before and after the intervention.
Change in Body Fat Mass | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Body fat mass measured by bioelectrical impedance analysis before and after the intervention.
Change in Body Mass Index | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Body mass index calculated as weight (kg) divided by height squared (m²) before and after the intervention.
Change in Percentage of Body Fat (% Body Fat) | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Percentage of total body fat assessed using bioelectrical impedance analysis before and after the intervention.
Change in Visceral Fat Level | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Visceral fat level measured using bioelectrical impedance analysis before and after the intervention.
Change in Extracellular Water | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Extracellular water assessed using bioelectrical impedance analysis before and after the intervention.
Change in Phase Angle | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Phase angle obtained through bioelectrical impedance analysis as an indicator of cellular health before and after the intervention.
Change in Waist Circumference | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Waist circumference measured with a flexible anthropometric tape at the midpoint between the last rib and the iliac crest before and after the intervention.
Change in Hip Circumference | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Hip circumference measured with a flexible anthropometric tape at the level of the greatest posterior protuberance of the buttocks before and after the intervention.
Change in Lower Body Functional Strength | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Lower body muscular strength assessed using the 30-second chair rise test before and after the intervention.
Change in Upper Body Strength | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Upper body muscular strength assessed using the arm curl test (both right and left arms) before and after the intervention.
Change in Functional Mobility, Dynamic balance and Risk of falls | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Functional mobility and dynamic balance assessed using the Timed Up and Go (TUG) test before and after the intervention.
Change in Static Balance | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Static balance assessed using the one-leg stand test (right and left legs) before and after the intervention.
Change in Upper Body Flexibility | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Upper body and shoulder flexibility assessed using the back scratch test for both right and left sides before and after the intervention.
Change in Squat Maximal Strength | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Maximal lower body strength assessed through the one-repetition maximum (1RM) squat test using a linear encoder before and after the intervention.
Change in Chest Press Maximal Strength | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Maximal upper body pushing strength assessed through the one-repetition maximum (1RM) chest press test using a linear encoder before and after the intervention.
Change in Incline Row Maximal Strength | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  Maximal upper body pulling strength assessed through the one-repetition maximum (1RM) incline row test using a linear encoder before and after the intervention.
Change in Squat Power | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  The power of lower body will be assessed through the squat exercise using a linear encoder before and after the intervention.
Change in Chess Press Power | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  The power of upper body will be assessed through the chess press exercise using a linear encoder before and after the intervention.
Change in Incline Row Power | Baseline, 1 month after surgery, 1 week before chemotherapy start, 1 week after chemotherapy completion, 6 months after surgery, and 5 months after initiation of endocrine/hormonal therapy.
  The power of upper body will be assessed through the incline row exercise using a linear encoder before and after the intervention.
Number of exercise sessions attended per participant in each exercise program | Throughout the intervention period
  Attendance rate to the supervised exercise sessions recorded throughout the intervention period.
Compliance With Prescribed Exercise Routines | Throughout the intervention period.
  Degree of compliance with the prescribed exercise program, including completion of assigned exercises, intensity, and volume.
Number of participants who dropout participation in each exercise program | Throughout the intervention period.
  Number of participants who discontinue participation in the exercise program before completing the intervention period.
Modification of the Prescribed Exercise Program | Throughout the intervention period
  Requirement for modifications to the prescribed exercise program due to clinical condition, treatment-related side effects, or physical limitations of the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- GOfit Vallerhermoso, Madrid, Madrid, Spain